CLINICAL TRIAL: NCT00004864
Title: A Phase I Open-Label Safety Study of Escalating Doses of Taxotere in Combination With Escalating Doses of GEM231 in Patients With Refractory Solid Tumors
Brief Title: Docetaxel and GEM 231 in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sridhar Mani, Prof. Dept of Medicine (Oncology), Montefiore Medical Center
Purpose: Treatment
Other Study IDs: CDR0000067520; P30CA013330 (NIH); AECM-1199906197; HYBRIDON-231-100A; NCI-G00-1666
Record Dates: First submitted 2000-03-07; First posted 2004-03-15 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — GEM231; Docetaxel

INTERVENTIONS:
Drug: GEM 231
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Gene therapy such as GEM 231 may inhibit the growth of cancer cells and make the tumor more sensitive to chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of combining docetaxel and GEM 231 in treating patients who have recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and maximum tolerated dose of docetaxel and GEM 231 in patients with recurrent or refractory solid tumors. II. Determine any preliminary antitumor activity of GEM 231 in this patient population.

OUTLINE: This is a dose escalation study of GEM 231 and docetaxel. Patients receive docetaxel IV over 1 hour on day 1, immediately followed by GEM 231 IV over 2 hours on days 1, 4, 8, and 11. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated with escalating doses of GEM 231 and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose limiting toxicity. Patients are followed monthly for 3 months.

PROJECTED ACCRUAL: A maximum of 1 patient will be accrued per week for this study until the maximum tolerated dose is reached.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor that is refractory to standard therapy or for which no standard therapy exists Measurable or evaluable disease No CNS metastases that are untreated, associated with seizures, or require intravenous medication and/or hospitalization

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.5 g/dL Hepatic: Bilirubin no greater than upper limit of normal (ULN), except Gilbert's syndrome PT and aPTT normal SGOT or SGPT less than 3 times ULN Renal: Creatinine less than 1.25 times ULN No renal tubular dysfunction (i.e., at least 2+ proteinuria within the past 2 weeks) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for 1 month prior to, during, and 3 months after study No other serious medical condition that would prevent compliance No serious infection Adequate venous access No known hypersensitivity to docetaxel or any oligodeoxynucleotides No prior peripheral neuropathy greater than grade 2 No psychological or geographical condition that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 week since prior transfusion Prior biologic therapy allowed and recovered No other concurrent biologic therapy Chemotherapy: Prior chemotherapy allowed and recovered No other concurrent chemotherapy Endocrine therapy: Prior hormonal therapy allowed and recovered Concurrent palliative hormonal therapy allowed Radiotherapy: Prior radiotherapy allowed and recovered No concurrent radiotherapy (except palliative) Surgery: At least 2 weeks since prior major surgery with wound complications Other: At least 2 weeks since prior investigational drugs No other investigational drugs during or within 28 days of study No concurrent CYP-3A metabolism dependent drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07 (Actual); Primary Completion 2000-06 (Actual); Study Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Comprehensive Cancer Center, The Bronx, New York, United States